CLINICAL TRIAL: NCT04003077
Title: Adjuvant Laser Meridian Massage in Heroin Addicts With Methadone Treatment: an Observational Case-controlled Study
Brief Title: Laser Meridian Massage in Heroin Addicts
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Ministry of Health and Welfare, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PMRPG8J0081; M08G1056 (Other Grant/Funding Number: Ministry of Health and Welfare); 201801823A3 (Other: Chang Gung Medical Foundation Institutional Review Board)
Record Dates: First submitted 2019-06-18; First posted 2019-07-01 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2019-06

CONDITIONS: Heroin Dependence
Keywords: Laser meridian massage; heroin addicts; methadone treatment; traditional Chinese medicine
MeSH Terms: conditions — Heroin Dependence

STUDY DESIGN:
Intervention Model Description: observational case-controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser meridian massage (Experimental): They are treated with laser meridian massage on the back including Bladder meridian and Governor vessel three times a week for 4 weeks.
  Interventions: Device: laser meridian massage
- Control (No Intervention): A control group of participants without laser meridian massage treatment are matched by age.

INTERVENTIONS:
Device: laser meridian massage — The participants will undergo 12 sessions of laser meridian massage, thrice a week, for 4 weeks, using a gallium aluminum arsenide LaserPen (maximal power, 150 mW; wavelength, 810nm; area of probe, 0.5cm^2; power density, 300mW/cm^2; pulsed wave; RJ-Laser, Reimers & Janssen GmbH, Waldkirch, Germany). The laser treatment will be applied to the back including Bladder meridian (BL11-25) and Governor vessel (GV3-14) for 15 minutes, to deliver a total treatment dose of 67.5J/cm^2.
  Arms: Laser meridian massage

SUMMARY:
A case-controlled study is conducted to investigate the effect of adjuvant laser meridian massage in heroin addicts with methadone treatment and establish the model of laser meridian massage treatment for drug addiction.

DETAILED DESCRIPTION:
Objective: To investigate the effect of adjuvant laser meridian massage in heroin addicts with methadone treatment and establish the model of laser meridian massage treatment for drug addiction.

Methods: A case-controlled study is conducted. Fifteen male heroin addicts are enrolled from Addiction Treatment Center as treatment group. They are treated with laser meridian massage on the back including Bladder meridian and Governor vessel three times a week for 4 weeks. A control group of participants without laser meridian massage treatment are matched by age. Check urine morphine before, 2 and 4 weeks of treatment. Subjects report their times or days of heroin use and self-fill Visual Analogue Scales of heroin craving / refusal of heroin use (0-10 points) during last week before, 2 and 4 weeks of treatment. Subjects report their quality of life using Short Form-12v2 before and 4 weeks of treatment. Obtain the subject's pulse diagnosis and heart rate variability after a single treatment. Independent t test, Mann-Whitney U test, chi-square test and Fisher's exact test were used to compare the differences between the treatment and control groups. Repeated measures ANOVA, Generalized estimating equations, paired t test and Wilcoxon Signed-Rank test were used for comparison between the treatment and control groups.

ELIGIBILITY:
Inclusion Criteria:

* Provide informed consent
* Male older than 20 years
* Diagnosed with opioid use disorder according to DSM-5 and received methadone treatment more than 1 month

Exclusion Criteria:

* Received Antidepressant or antipsychotic
* Received Chinese herb or acupuncture treatment during last 30 days
* Critical illness
* Did not meet the physician's assessment for recruitment
* Patients with Human immunodeficiency virus infection
* Did not provide informed consent

Ages: 20 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-02-26 (Actual); Primary Completion 2020-04-16 (Estimated); Study Completion 2020-04-16 (Estimated)

PRIMARY OUTCOMES:
Heroin use | 2 weeks of treatment
  Times or days of heroin use during last week
Heroin use | 4 weeks of treatment
  Times or days of heroin use during last week
Urine morphine | 2 weeks of treatment
  Obtainurinary morphine concentration
Urine morphine | 4 weeks of treatment
  Obtain urinary morphine concentration

SECONDARY OUTCOMES:
Heroin craving / refusal of heroin use | 2 weeks of treatment
  Obtain Visual Analogue Scales (VAS) of heroin craving / refusal of heroin use (0-10 points) during last week. VAS score 0 of heroin craving indicates no heroin craving, while VAS 10 indicates strongest heroin craving. VAS 0 of refusal of heroin use indicates no refusal of heroin, while VAS 10 indicates absolute refusal of heroin.
Heroin craving / refusal of heroin use | 4 weeks of treatment
  Obtain Visual Analogue Scales (VAS) of heroin craving / refusal of heroin use (0-10 points) during last week. VAS score 0 of heroin craving indicates no heroin craving, while VAS 10 indicates strongest heroin craving. VAS 0 of refusal of heroin use indicates no refusal of heroin, while VAS 10 indicates absolute refusal of heroin.
Short Form-12v2 Health Survey | 4 weeks of treatment
  The SF-12v2® Health Survey (SF-12v2) is a multipurpose, short-form health survey with 12 questions that yields an eight-scale proﬁle of functional health and well-being, as well as two psychometrically based physical and mental health summary measures and a preference-based health utility index.
  The PRO CoRE, part of the Smart Measurement® System suite of products and Optum's upgrade to the QualityMetric Health Outcomes™ Scoring Software, is used for scoring the SF-12v2® Health Survey.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hu WL, Tsai MC, Kuo CE, Liu CT, Wu SY, Wu TC, Hung YC. Adjuvant laser meridian massage in men with opioid use disorder on methadone maintenance treatment: Protocol for a case-controlled study. Medicine (Baltimore). 2019 Sep;98(39):e17319. doi: 10.1097/MD.0000000000017319. PMID 31574863